CLINICAL TRIAL: NCT00581945
Title: A Randomized, Double-blind, Placebo Controlled, Exploratory Study to Assess the Safety and Efficacy of Multiple Doses of ACZ885 in Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: Safety and Efficacy of Multiple Doses of Canakinumab (ACZ885) in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CACZ885B2204
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canakinumab (Experimental): Participants received an initial dose of 1 mg/kg canakinumab (ACZ885) via intravenous infusion. Four weeks later, participants received a dose of 3 mg/kg canakinumab, and another dose of 3 mg/kg two weeks later. Thereafter, participants received doses of 6 mg/kg every four weeks until completion of the 45-week treatment period.
  Interventions: Drug: Canakinumab
- Placebo (Placebo Comparator): Participants received a matching placebo intravenous infusion at weeks 1, 5, 7, and thereafter every four weeks until completion of the 45-week treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab — The dose of canakinumab (ACZ885) administered was individualized, based on the subject's weight pre-dose, and was administered via intravenous infusion.
  Arms: Canakinumab
Drug: Placebo — Matching placebo to ACZ885 administered via intravenous infusion.
  Arms: Placebo

SUMMARY:
Was to evaluate the safety, tolerability and efficacy of multiple doses of canakinumab (ACZ885) vs. placebo when administered via intravenous infusion (IV), on pulmonary function in patients with COPD

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects from 40-80 years (inclusive) of age
* Subjects have a clinical diagnosis of COPD
* Smokers or Ex-smokers with a smoking history of at least 20 pack years
* Post-bronchodilator forced expiratory volume in 1 second (FEV1 ) at screening ≤ 50% of the predicted normal value
* Post-bronchodilator FEV1/FVC ratio < 70%
* History of at least one treated exacerbation during the 24 months year prior to screening or C-Reactive Protein (CRP) ≥3.47 mg/L,
* Subjects should have no concomitant other lung disease or significant concomitant medical conditions that would affect the subjects' safety when participating in the study, or that would be expected to impact on the results of the study
* Female subjects must have been surgically sterilized at least 6 months prior to screening or must be using two forms of contraception, or postmenopausal women
* Able to provide written informed consent prior to study participation.
* Able to communicate well with the investigator and comply with the requirements of the study.

Exclusion Criteria:

* COPD exacerbation(s) requiring treatment within 4 weeks prior to first dosing
* History of lung reduction surgery
* Any undiagnosed nodule on chest x-ray
* Presence of certain medical conditions as specified by the protocol
* Subjects requiring oral or parenteral corticosteroids equivalent to > 10 mg/day or > 20 mg every other day of prednisone or prednisolone
* Documented homozygous alpha-1 antitrypsin deficiency.
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing.
* A past medical history of clinically significant electrocardiogram (ECG) abnormalities or a family history of a prolonged QT-interval syndrome.
* A known hypersensitivity to drugs similar to the study drug.
* History of immunocompromise, including a positive HIV test result.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* History of drug or alcohol abuse within the 12 months prior to screening or evidence of such abuse as indicated by the laboratory assays conducted during screening.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2007-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NOVARTIS, Principal Investigator — Novartis investigator site
Locations (11):
- United States (11):
  - Novartis Investigator Site, Anaheim, California
  - Novartis Investigator Site, Los Angeles, California
  - Novartis Investigator Site, Panama City, Florida
  - Novartis Investigator Site, Marietta, Georgia
  - Novartis Investigator Site, Baltimore, Maryland
  - Novartis Investigator Site, Livonia, Michigan
  - Novartis Investigator Site, Minneapolis, Minnesota
  - Novartis Investigator Site, Omaha, Nebraska
  - Novartis Investigator Site, Buffalo, New York
  - Novartis Investigator Site, Spartanburg, South Carolina
  - Novartis Investigator Site, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Canakinumab: Participants received an initial dose of 1 mg/kg canakinumab via intravenous infusion. Four weeks later, participants received a dose of 3 mg/kg canakinumab, and another dose of 3 mg/kg two weeks later. Thereafter, participants received doses of 6 mg/kg every four weeks until completion of the 45-week treatment period.
Period: Overall Study
Arm/Group | Canakinumab | Placebo
Started | 74 | 73
Completed | 65 | 63
Not Completed | 9 | 10
Not completed — Adverse Event | 4 | 4
Not completed — Unsatisfactory therapeutic effect | 2 | 0
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab | Placebo | Total
Number analyzed (Participants) | 74 | 73 | 147
Age Continuous [Mean (Standard Deviation); unit: years] | 63.9 (7.70) | 63.6 (7.92) | 63.7 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 31 | 59
  Male | 46 | 42 | 88

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: Forced expiratory volume in 1 second (FEV1) is the amount of air that can be exhaled in one second. FEV1 was measured by spirometry performed at approximately the same time of day on each visit to avoid diurnal variation. All spirometry calibrations and evaluations followed the recommendations of the American Thoracic Society / European Respiratory Society guidelines for acceptability. A positive change from baseline in FEV1 indicates improvement in lung function.
Time Frame: Baseline, Week 25 and Week 45
Population: The safety population consisted of all randomized patients who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 74 | 73
Liters
  Change from Baseline at Week 25 | -0.027 (0.1725) | -0.006 (0.2545)
  Change from Baseline at Week 45 | -0.044 (0.1542) | -0.033 (0.2512)

2. Secondary Outcome: Number of Participants Who Experienced Serious Adverse Events or Discontinued Due to Adverse Events
Description: Safety was assessed by the number of participants with serious adverse events and/or adverse events leading to study discontinuation. A summary of adverse events is presented with this outcome, additional details are provided in the Adverse Events section.
Time Frame: Adverse events were collected during the 45 week treatment period and the 12 week follow-up period.
Population: The safety population consisted of all randomized patients who received at least one dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 74 | 73
Participants
  Serious Adverse Events | 23 | 14
  Death | 1 | 0
  Discontinued due to Adverse Events | 4 | 4
  Discontinued due to Serious Adverse Events | 3 | 4
  Discontinued due to non-serious AEs | 1 | 0

3. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second Percent Predicted
Description: The FEV1 percent predicted expresses FEV1 as a percentage of the "predicted values" for participants of similar characteristics (height, age, sex, and sometimes race and weight). A positive change from baseline in FEV1 % predicted indicates improvement in lung function.
Time Frame: Baseline, Week 25 and Week 45
Population: Safety population
Measure: Mean (Standard Deviation); unit: Percent of predicted
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 74 | 73
Percent of predicted
  Change from Baseline at Week 25 | -0.2 (6.42) | 0.3 (8.86)
  Change from Baseline at Week 45 | -1.0 (5.35) | -0.7 (8.49)

4. Primary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: Forced Vital Capacity is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC was assessed by spirometry. A positive change from baseline in FVC indicates improvement in lung function.
Time Frame: Baseline, Week 25 and Week 45
Population: Safety population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 74 | 73
liters
  Change from Baseline at Week 25 | -0.010 (0.3720) | -0.061 (0.4856)
  Change from Baseline at Week 45 | -0.039 (0.3122) | -0.065 (0.5170)

5. Primary Outcome: Change From Baseline in Slow Vital Capacity (SVC)
Description: Vital Capacity is the amount of air that can be forcibly exhaled from the lungs after a full inhalation. Slow Vital Capacity (SVC) test is performed by having the patient slowly and completely blow out all of the air from their lungs. A positive change from baseline in SVC indicates improvement in lung function.
Time Frame: Baseline, Week 25 and Week 45
Population: Safety population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 74 | 73
liters
  Change from Baseline at Week 25 | -0.029 (0.3746) | -0.019 (0.5082)
  Change from Baseline at Week 45 | -0.062 (0.3727) | -0.017 (0.5379)

6. Primary Outcome: Change From Baseline in Forced Expiratory Flow 25% to 75%
Description: The forced expiratory flow (FEF) 25%-75% measurement describes the amount of air expelled from the lungs during the middle half (25% - 75%) of the forced vital capacity test and is measured using spirometry. A positive change from baseline in FEF indicates improvement in lung function.
Time Frame: Baseline, Week 25 and Week 45
Population: Safety population
Measure: Mean (Standard Deviation); unit: L/sec
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 74 | 73
L/sec
  Change from Baseline at Week 25 | -0.022 (0.1060) | -0.002 (0.1111)
  Change from Baseline at Week 45 | -0.024 (0.0898) | -0.012 (0.1244)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 45-week treatment period.
Arm/Group | Canakinumab | Placebo
Serious Adverse Events (participants affected / at risk) | 23/74 | 14/73
Other Adverse Events (participants affected / at risk) | 59/74 | 51/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=74) | Placebo (N=73)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 1
Oral allergy syndrome (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 3
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=74) | Placebo (N=73)
Diarrhoea (Gastrointestinal disorders) | 5 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 5 | 6
Vomiting (Gastrointestinal disorders) | 5 | 1
Pyrexia (General disorders) | 7 | 7
Candidiasis (Infections and infestations) | 2 | 4
Gastroenteritis viral (Infections and infestations) | 4 | 2
Oral candidiasis (Infections and infestations) | 3 | 4
Sinusitis (Infections and infestations) | 6 | 5
Upper respiratory tract infection (Infections and infestations) | 9 | 4
Urinary tract infection (Infections and infestations) | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 38 | 36
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Hypertension (Vascular disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.